CLINICAL TRIAL: NCT00328900
Title: Measurement of Stress During Anesthesia With "Pain Detector" on Patients Receiving Atropine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rikshospitalet University Hospital (Other)
Responsible Party: Hanne Storm MD.PhD, Rikshospitalet, UIO
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: S-03113
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2007-04

CONDITIONS: Hemorrhoids; Fissure in Ano
Keywords: Galvanic skin response; Anesthesia; Atropine
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Administration of 0,7 mg of atropine
Device: Measurement of skin conductance with Pain detector

SUMMARY:
24 patients randomly divided into two groups, one of the groups receiving atropine in addition to the planned anaesthesia. Skin conductance parameters to be compared between the two groups.

DETAILED DESCRIPTION:
Skin conductance (SC), in terms of numbers of skin conduction fluctuations (NSCF), amplitude and mean skin conductance level, reflect the activity in the sympathetic postganglionic cholinergic fibers which innervate the palmar and plantar sweat glands. Skin conductance, especially numbers of skin conductance fluctuations, may be a promising tool to monitor anesthesia. Atropine, an anticholinergic agent, acts as an antagonist on the muscarinic receptors of the sweat glands and inhibits their secretion in a dose-dependent way. The aim of this study was to find out to what degree SC is influenced by i.v. administration of atropine.

Study hypothesis: SC is not influenced by i.v. administration of atropine.

ELIGIBILITY:
Inclusion Criteria:

* Patients in ASA-group 1-2
* Operations (anal fissures, anal fistulas and haemorrhoids) lasting for less than one hour
* informed consent
* BMI <30

Exclusion Criteria:

* Patients using any medication known to influence the autonomous nervous system
* Patients with contraindications to atropine (e.i. fibrillation, glaucoma ect)
* BMI >30
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Number of skin conductance fluctuations

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Storm, PhD, Study Director — Rikshospitalet University Hospital
Locations (1):
- Ulleval University Hospital, Oslo, Norway